CLINICAL TRIAL: NCT04672759
Title: A Real-world Study of Consolidation Durvalumab for Stage III Unresectable Non-small Cell Lung Cancer in China and Safety Data on Durvalumab in Chinese Patients With Lung Cancer（PACIFIC-PUMCH-R）
Brief Title: A Real-world Study of Durvalumab for Lung Cancer in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Li Zhang, Chief Physician, Peking Union Medical College Hospital
Other Study IDs: PACIFIC-PUMCH-R
Record Dates: First submitted 2020-12-07; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Non Small Cell Lung Cancer Stage III; Small-Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — durvalumab; Drug Therapy; Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Cohort 1 will include patients with unresectable stage III non-small cell lung cancer. Patients receive durvalumab as an intravenous infusion over 60 minutes on day 1. Courses repeat every 21 days for up to 12 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Durvalumab
- Cohort 2: Cohort 2 will enroll patients with histologically or cytologically confirmed NSCLC or SCLC who will or have received chemotherapy/radiotherapy at the physician's discretion.
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — Patients receive durvalumab as an intravenous infusion over 60 minutes on day 1. Courses repeat every 21 days for up to 12 months in the absence of disease progression or unacceptable toxicity.
Drug: Durvalumab — Durvalumab monotherapy or combined with chemotherapy and/or radiotherapy.
  Other Names: chemotherapy, radiotherapy

SUMMARY:
PACIFIC-PUMCH-R is an ambispective cohort study that will enroll approximately 100 patients with lung cancer who have received at least one dose of durvalumab between July 2020 and July 2021. Patient selection and data collection will be from Peking Union Medical College Hospital.

Cohort 1 will include patients with unresectable stage III non-small cell lung cancer (according to the Staging Manual in Thoracic Oncology, version 7, of the International Association for the Study of Lung Cancer) who did not have disease progression after concurrent chemoradiotherapy. The primary objective of Cohort 1 is to assess the effectiveness of durvalumab in a real-life setting by evaluating PFS and OS in Chinese patients.

Cohort 2 will enroll patients with histologically or cytologically confirmed NSCLC or SCLC who have received chemotherapy/radiotherapy at the physician's discretion. And this Cohort aimed to assess the safety of durvalumab for the treatment of lung cancer in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Patient capable of proper therapeutic compliance, and accessible to correct follow-up.
2. Written Informed Consent (IC) for trial treatment must be signed and dated by the patient and the investigator prior to any trial-related evaluation and/or intervention.
3. Age ≥ 18 years at time of study entry or adult according to each country regulations for age of majority.
4. Patients must have histologically or cytologically documented diagnosis of NSCLC with a locally advanced, or locally recurrent, unresectable (stage III) disease (according to American Joint Committee on Cancer [AJCC] lung cancer edition 8). Histologically or cytologically documented extensive disease (American Joint Committee on Cancer Stage (8th edition) IV SCLC. Brain MRI or high-quality brain CT with intravenous contrast at the time of staging mandatory is strongly recommended.
5. Patients who received definitive concurrent chemoradiation therapy and have not progressed were enrolled in the Cohort 1. Patients who received chemotherapy, radiotherapy or sequential chemotherapy were enrolled in the Cohort 2.
6. Tumour sample requirements: Provision of an unstained tumor samples in a quantity sufficient to allow for analysis (≤3 months newly collected sample is preferred, ≤6 months archival sample is also accepted.)
7. No prior exposure to immune-mediated therapy including, but not limited to, other.
8. anti-CTLA-4, anti-PD-1, anti-PD-L1, and anti-programmed cell death ligand 2.
9. (anti-PD-L2) antibodies, excluding therapeutic anticancer vaccines.

Exclusion Criteria:

1. Patients should not enter the study if any of the following exclusion criteria are fulfilled:
2. History of allogenic organ transplantation.
3. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis with the exception of diverticulosis, systemic lupus erythematosus, sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, and uveitis, etc]). The following are exceptions to this criterion:

   * Patients with vitiligo or alopecia
   * Patients with hypothyroidism (eg, following Hashimoto syndrome) and stable
   * on hormone replacement
   * Any chronic skin condition that does not require systemic therapy
   * Patients without active disease in the last 5 years may be included but only after
   * consultation with the Study Physician
   * Patients with celiac disease controlled by diet alone
4. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, interstitial lung disease, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
5. History of another primary malignancy except for

   * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence
   * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
   * Adequately treated carcinoma in situ without evidence of disease
6. History of active primary immunodeficiency.
7. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen [HbsAg] result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HbsAg) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
8. Mixed small cell and non-small cell lung cancer histology
9. Any unresolved toxicity CTCAE ≥Grade 2 from the prior chemoradiation therapy. Patients with irreversible toxicity that is not reasonably expected to be exacerbated by study drug may be included (eg, hearing loss) after consultation with the AstraZeneca/MedImmune medical monitor.
10. Patients with ≥Grade 2 pneumonitis from prior chemoradiation therapy
11. Known allergy or hypersensitivity to durvalumab or any of their excipients
12. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment
13. Receipt of live, attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
14. Recent major surgery within 4 weeks prior to entry into the study (excluding the placement of vascular access) that would prevent administration of study drug
15. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids or local steroid injections (eg, intra articular injection).
    * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent.
    * Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication). Premedication with steroids for chemotherapy is acceptable. Systemic steroid administration required to manage toxicities arising from radiation therapy delivered as part of the chemoradiation therapy for locally advanced NSCLC is allowed
16. Participation in another clinical study with an IP during the last 4 weeks
17. Previous enrolment or randomisation in the present study
18. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
19. Prior randomization or treatment in a previous durvalumab and/or tremelimumab clinical study regardless of treatment arm assignment.
20. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from Screening to 90 days after the last dose of durvalumab monotherapy
21. According to the investigator, if the subject is unable to comply with procedures required by the clinical investigation, the subject is not allowed to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will enroll approximately 100 patients with lung cancer who have received at least one dose of durvalumab between July 2020 and July 2022. Patient selection and data collection will be from Peking Union Medical College Hospital.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-07-28 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (Cohort 1) | Tumor scans performed at baseline then every ~8 weeks up to 48 weeks, then every ~12 weeks thereafter until confirmed disease progression. Assessed up to a maximum of approximately 3 years
  PFS is defined as time from the index date (date of the first dose of durvalumab) to the date of the first documentation of progressive disease (PD) or death from any cause, whichever occurs first. Per RECIST 1.1 modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions is also considered PD.
Overall Survival (Cohort 1) | From baseline until death due to any cause. Assessed up to a maximum of approximately 4 years.
  OS is defined as the time from randomization to the time of death from any cause.
Number of Participants With one or more Adverse Events (Cohort 2) | Baseline until up to 90 days after end of treatment.
  Adverse events (AE) are graded using the Common Terminology Criteria for Adverse Events (CTCAE) v4.0. Grade refers to the severity of the AE. The CTCAE v4.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE.

SECONDARY OUTCOMES:
Objective response rate (Cohort 1) | Tumor scans performed at baseline then every ~8 weeks up to 48 weeks, then every ~12 weeks thereafter until confirmed disease progression. Assessed up to a maximum of approximately 4 years.
  Objective response is defined as best overall response (CR or PR) across all assessment timepoints during the period from enrolment to termination of trial treatment.
Duration of Response (Cohort 1) | Tumor scans performed at baseline then every ~8 weeks up to 48 weeks, then every ~12 weeks thereafter until confirmed disease progression. Assessed up to a maximum of approximately 4 years.
  For participants who demonstrated CR or PR, DOR is defined as the time from the first documented evidence of CR or PR until PD or death from any cause, whichever occurs first. Per RECIST 1.1 modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ, or death from any cause, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm.
Time to death or distant metastasis (Cohort 1) | Tumor scans performed at baseline then every ~8 weeks up to 48 weeks, then every ~12 weeks thereafter until confirmed disease progression. Assessed up to a maximum of approximately 4 years.
  TTDM will be defined as the time from the index date (date of the first dose of durvalumab) to the first date of distant metastasis or death in the absence of distant metastasis.
Time from the index date to second progression (Cohort 1) | Following confirmed progression, patients were assessed every ~12 weeks until second disease progression. Assessed up to a maximum of approximately 4 years.
  PFS2 will be defined as the time from the index date to the earliest of the progression event subsequent to that used for the PFS endpoint or death.
Number of Participants With one or more Adverse Events (Cohort 1) | Baseline until up to 90 days after end of treatment.
  Adverse events (AE) are graded using the Common Terminology Criteria for Adverse Events (CTCAE) v4.0. Grade refers to the severity of the AE.
Change from Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Global Health Status/Quality of Life | At baseline, every 4 weeks for first 8 weeks, then every ~8 weeks until 48 weeks, then every ~12 weeks thereafter until confirmed disease progression. Assessed up to a maximum of approximately 4 years.
  The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. The EORTC Quality of Life Questionnaire and Lung Cancer Module 13 (QLQ-LC13) is a supplemental lung cancer-specific module used in combination with QLQ-C30. An increase in combined score indicates improvement in quality of life.
Progression-free Survival (Cohort 2) | Tumor scans performed at baseline then every ~8 weeks up to 48 weeks, then every ~12 weeks thereafter until confirmed disease progression. Assessed up to a maximum of approximately 3 years.
  PFS is defined as time from the index date (date of the first dose of durvalumab) to the date of the first documentation of progressive disease (PD) or death from any cause, whichever occurs first. Per RECIST 1.1 modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions is also considered PD.
Overall Survival (Cohort 2) | From baseline until death due to any cause. Assessed up to a maximum of approximately 4 years.
  OS is defined as the time from randomization to the time of death from any cause.
Objective response rate (Cohort 2) | Tumor scans performed at baseline then every ~8 weeks up to 48 weeks, then every ~12 weeks thereafter until confirmed disease progression. Assessed up to a maximum of approximately 4 years.
  Objective response is defined as best overall response (CR or PR) across all assessment timepoints during the period from enrolment to termination of trial treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No